CLINICAL TRIAL: NCT07256028
Title: Use of Stable Isotopic Dilution to Assess the Bioavailability of Indispensable Amino Acids in Children With Environmental Enteropathy Dysfunction (IAA-EED)
Brief Title: Indispensable Amino Acids Bioavailability in Children With Environmental Enteropathy Dysfunction (IAA-EED)
Acronym: IAA-EED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morocco's National Centre for Energy, Sciences and Nuclear Techniques (Other)
Collaborators: CCTD, Centre Hospitalier Ibn Sina,Morocco (Unknown); AgroParisTech (Other)
Responsible Party: Principal Investigator, Mohammed El Mzibri, Head of the Life Sciences Division, Morocco's National Centre for Energy, Sciences and Nuclear Techniques
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IAEA Research Contract 24437
Record Dates: First submitted 2025-11-17; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Environmental Enteric Dysfunction
Keywords: Indispensable amino acids; Environmental enteric dysfunction; bioavailability; amino acids supplementatuion

STUDY DESIGN:
Intervention Model Description: The 18-36-month-old children in the intervention arm will receive milk with IAA supplementation for 28 days, while children in the control group will receive only milk for the same duration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm with IAA supplemntation (Experimental): 18-36-month-old children will receive daily 100 ml of milk supplemented with IAA
  Interventions: Dietary Supplement: Indispensable amino acids supplemntation
- Arm without IAA supplementation (Experimental): 18-36 months-aged children will receive only milk
  Interventions: Dietary Supplement: Without Indispensable amino acids supplementation

INTERVENTIONS:
Dietary Supplement: Indispensable amino acids supplemntation — 18-36-month-old children in the intervention arm will receive milk with IAA supplementation for 28 days, while children in the control group will receive only milk for the same duration
  Arms: Arm with IAA supplemntation
Dietary Supplement: Without Indispensable amino acids supplementation — 18-36-month-old children in the intervention arm will receive milk with IAA supplementation for 28 days, while children in the control group will receive milk without IAA during the same duration
  Other Names: IAA supplemntation
  Arms: Arm without IAA supplementation

SUMMARY:
In Morocco, large efforts have been made to enhance nutritional status and health conditions of children. Accordingly, stunting was reduced and the prevalence of stunting have decreased from 28,6% in 1987 to 14,9% in 2011. Many factors, including improved nutrition, have influenced this decrease, and are reinforced to maintain this low prevalence of stunting. Of interest, quality diet, specifically with reference to its protein quality, has contributed to improve the nutritional status of the Moroccan population. However, infectious diseases are still important and in some areas many children are of high risk to develop EED that alter intestinal permeability and microbial translocation, and lead to systemic inflammation. During childhood, protein supply is of a great interest and indigestibility of these proteins and/or malabsorption of indispensable amino acids will affect children growth and many physiological and cognitive functions. This project was planned to assess indispensable amino acids during EED and to to assess the impact of some interventions (amino acids supplementation / medical treatment) on the nutritional status of children.

This study will be carried out according to a trilogy of close collaboration between CNESTEN, Pr Claire Gaudichon from AgroParisTech (France) who will provide technical assistance and scientific accompaniment during the progress of the project, she will also participate in the data analysis, exploitation and valorization of results and the department of Pediatric Hepatology Gastroenterology and Nutrition-P III at the Children's Hospital in Rabat.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial to determine if indispensable amino acid (IAA) supplementation can improve intestinal barrier dysfunction in Moroccan patients aged 18-36-month-old with stunting or severe stunting. The primary endpoint will be change in gut permeability as assessed by the lactulose/rhamnose (LR) ratio, while secondary endpoint will focus on change in amino acid absorption using an isotope tracer test. IAA supplementation will be given daily for 28 days, and evaluation of the major endpoints will be at baseline and 28 days

ELIGIBILITY:
Inclusion Criteria:

* Stunting estimated at least - 2 z score height -for-age
* Abnormal intestinal morphology on jejunal biopsy showing features for EED:
* mucosal inflammation,
* villous blunting
* altered barrier integrity

Exclusion Criteria:

* Celiac disease
* Presence of anti-tissue transglutaminase antibodies.
* Primary immunodeficiency disorders
* Inflammatory bowel disease
* Intestinal inflammation food allergy

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Use of the lactulose/rhamnose (LR) ratio to assess improvement in gut permeability among stunted Moroccan children aged 18-36 months after 28 days of Indispensable Amino Acids (IAA) supplementation. | The procedure involves assessing gut permeability at enrolment and again after 28 days of IAA supplementation.
  The purpose of this measure is to assess gut permeability efficiency and whether supplementation with IAA can improve it. In fact, the lactulose/rhamnose (LR) ratio or the dual-sugar test is a non-invasive test used to measure intestinal permeability. It works by orally administering of two inert sugar molecules, lactulose and rhamnose, then measuring their excretion in urine; a higher LR ratio suggests increased intestinal permeability, often indicating damage to the gut lining. This test is useful in research and clinical settings for assessing conditions that affect the small intestine.
Use of Dual-Stable Isotope Test (DSIT) to assess improvement of the true ileal bioavailability of IAA among stunted Moroccan children aged 18-36 months after 28 days of IAA supplementation. | The procedure involves assessing the rate of IAA bioavailability at enrolment and again after 28 days of IAA supplementation.
  The purpose of this measure is to assess the rate of IAA bioavailability and determine whether IAA supplementation can improve it. To this end, the Dual-Stable Isotope Test (DSIT) will be used. The DSIT is a minimally invasive method for measuring the true ileal bioavailability of IAAs in humans, using a meal containing both the 2H-labeled test protein and the 13C-labeled reference protein. In this study, children will consume a test meal (milk) containing both the 2H-AA mix (1.25 mg/kg body weight) and the U-13C spirulina (10 mg/kg body weight). To carry out this technique, two blood (plasma) samples will be collected, one before the meal is administrated and the second 5hours after afterwards. A portion of the meal will be frozen at -80°C for later analysis of the two isotopes. The bioavailability of each IAA is calculated by comparing the ratio of the two isotopes in the plasma samples to their ratio in the original test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El Mzibri, Principal Investigator — Centre National de l'Energie, des Sciences et des Techniques Nucléaire; Toufik Meskini, Professor, Study Director — Department of Pediatric Hepatology Gastroenterology and Nutrition-P III. Children's hospital of Rabat - the Ibn Sina University Hospital Center
Locations (1):
- department of Pediatric Hepatology Gastroenterology and Nutrition-P III. Children's hospital of Rabat - the Ibn Sina University Hospital Center, Rabat, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No
Only scientific results will be published